CLINICAL TRIAL: NCT04060264
Title: Randomized, Open-Label, International, Multi-center, Comparative Study of Efficacy and Safety of BCD-148 (JSC BIOCAD, Russia) and Soliris® in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Clinical Trial of BCD-148 and Soliris® for the Treatment of Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-148-2
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: During the main period (first 27 weeks), test product BCD-148 and reference product Soliris®.
  After Week 27, patients of both study arms will be switched to BCD-148 900 mg biweekly as maintenance therapy. Duration of this maintenance therapy will be 25 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-148 (Experimental): 14 participants in BCD-148 group. During the main period (first 27 weeks), test product BCD-148 will be administered as 25- to 45-minute intravenous infusions.
  After Week 27 BCD-148 900 mg will be administered biweekly as maintenance therapy.
  Interventions: Biological: BCD-148
- Soliris (Active Comparator): 14 participants in Soliris group. During the main period (first 27 weeks), Soliris® will be administered as 25- to 45-minute intravenous infusions.
  After Week 27, patients be switched to BCD-148 900 mg biweekly as maintenance therapy.
  Interventions: Biological: BCD-148; Biological: Soliris

INTERVENTIONS:
Biological: BCD-148 — Active substance of BCD-148 is eculizumab - a monoclonal antibody that targets complement protein C5.
  Cycle 1 (induction therapy): 600 mg of eculizumab QW for the first four weeks; Cycle 2 (maintenance therapy): 900 mg of eculizumab at Week 5 and 900 mg of eculizumab every 14±2 days until Week 27 (inclusive) afterwards (dosing regimen for the main study period).
  QW - once weekly
Biological: Soliris — Active substance of Soliris is eculizumab - a monoclonal antibody that targets complement protein C5.
  Cycle 1 (induction therapy): 600 mg of eculizumab QW for the first four weeks; Cycle 2 (maintenance therapy): 900 mg of eculizumab at Week 5 and 900 mg of eculizumab every 14±2 days until Week 27 (inclusive) afterwards (dosing regimen for the main study period).
  Arms: Soliris

SUMMARY:
This clinical study is a randomized, open-label, international, multi-center, comparative study of efficacy and safety of BCD-148 and Soliris® in PNH patients.

It is planned to investigate the efficacy, safety, and immunogenicity of one-year eculizumab course in this study.

PNH - Paroxysmal nocturnal hemoglobinuria

ELIGIBILITY:
Inclusion Criteria:

1. He/she gave written informed consent.
2. Male or female ≥18 and ≤65 years of age.
3. PNH diagnosis documented by flow cytometry data at screening .
4. PNH granulocyte clone size ≥10% (according to flow cytometry performed at screening).
5. Lactate dehydrogenase (LDH) level ≥1.5 times the upper limit of normal (ULN) at screening and at least one of the following symptoms/syndromes: hemoglobinuria, thrombotic complications, transfusion-dependent chronic hemolysis, anemic syndrome, acute kidney injury episodes or chronic kidney disease, pulmonary hypertension, and signs of smooth muscle dystonia (e.g., abdominal pain, dysphagia, erectile dysfunction, and etc.) within three months before informed consent.
6. Platelet count ≥30х109/L at screening.
7. Absolute count of neutrophil granulocytes ≥0.75х109/L at screening.
8. Willingness to undergo vaccination against Neisseria meningitidis during the screening period and at least 14 days before the first administration of an investigational product .
9. If immunosuppressive drug products are used, the duration of this therapy should be at least three months by informed consent date.
10. The willingness of patients and their sexual partners of childbearing potential to use reliable contraception methods starting from the informed consent, throughout the study, and for four weeks after the last dose of an investigational product. This requirement does not apply to patients who underwent surgical sterilization and women with menopause established more than two years ago. Reliable contraception methods include one barrier method in combination with one of the following: spermicides or an intrauterine device.
11. The patient is able, in the Investigator's opinion, to follow study procedures.

Exclusion Criteria:

1. History of meningococcal infection (either well-documented or according to oral information provided by a patient).
2. Other well-documented complement deficiencies (except for those concerning complement component 5).
3. History of bone marrow transplantation (either well-documented or according to oral information provided by a patient).
4. HIV, hepatitis B, active hepatitis C, and syphilis .
5. A patient with newly diagnosed or relapsing aplastic anemia and/or progressive bone marrow failure with indications for allogeneic bone marrow transplantation or combined immunosuppressive therapy within 6 months after informed consent.
6. Acute infection (either well-documented and/or according to oral information provided by a patient) within 4 weeks before informed consent and/or during the screening period and/or relapse of chronic disease at the moment of informed consent and/or during the screening period .
7. Any other chronic diseases present at the time of the informed consent which can negatively affect the patient's safety during the study, in the Investigator' opinion.
8. Use of eculizumab and/other anti-C5 monoclonal antibodies within three months before informed consent .
9. Hypersensitivity to any of BCD-148/Soliris® ingredients, murine proteins and other ingredients of these drug products, and to any of meningococcal vaccine ingredients.
10. Documented malignancy, except for cured basal cell carcinoma or cervical carcinoma in situ .
11. A known alcoholic or drug abuse or signs of present alcoholic/drug abuse that, in the Investigator's opinion, can be a contraindication to treatment with an investigational product or limit treatment compliance.
12. Participation in other clinical studies within 30 days before informed consent and during this study.
13. Pregnancy or lactation or planning for pregnancy/paternity during the clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
AUC LDH | Weeks 5-27
  AUC - Area Under Curve of Lactate dehydrogenase

SECONDARY OUTCOMES:
The proportion of patients with thrombotic complications | week 27, week 52
The proportion of patients who required red blood cell transfusion | week 27, week 52
The proportion of patients with stable Hb level during the maintenance therapy period | Weeks 5-27
Mean Hb level over the maintenance therapy period | Weeks 5-27
Frequency of breakthrough hemolysis episodes | week 27, week 52
Changes in LDH level over time | week 27, week 52
Change in the count of circulating red blood cells with the PNH phenotype RBC | week 27, week 52
  Red blood cells (RBC )
Change in mean FACIT-Fatigue score | week 27, week 52
  FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
Change in mean EORTC QLQ-C30 score | week 27, week 52
  EORTC QLQ-C30 is questionnaire developed to assess the quality of life. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
  QLQ - Quality of Life Questionnaire
The proportion of patients with AE/SAE related to an investigational product, in the Investigator's opinion | week 27, week 52
  AE - adverse event, SAE - serious adverse event
The proportion of patients with СТСАЕ v.5.0 Grade 3-4 AE related to an investigational product, in the Investigator's opinion, by arm | week 27, week 52
The proportion of patients who discontinued early due to AE/SAE related to an investigational product, in the Investigator's opinion, by arm | week 27, week 52
The proportion of BAb- and NAb-positive patients. | week 27, week 52
  BAb - Binding antibodies, NAb - neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JSC BIOCAD
Locations (1):
- Federal State Budgetary Educational Institution of Higher Education "Academician I.P. Pavlov First St. Petersburg State Medical University" of the Ministry of Healthcare of Russian Federation, Saint Petersburg, Russia